CLINICAL TRIAL: NCT00957177
Title: Effect of Preoperative Pregabalin Administration on the Postoperative Opioid Consumption in Patients Undergoing Nephrectomy
Brief Title: Analgetic Effect of Preoperative Pregabalin in Patients Undergoing Nephrectomy
Acronym: PregabaNeph
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sandner-Kiesling Andreas, Prof. Dr., Medical Universitiy of Graz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PregabaNeph
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Pregabalin group (Active Comparator): Receiving 300mg pregabalin preoperative
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — 300mg pregabalin orally 1 hour before operation
  Other Names: Lyrica
  Arms: Pregabalin group
Drug: Placebo — Placebo
  Other Names: Control
  Arms: Placebo

SUMMARY:
Pregabalin 300mg or placebo are administered 1 hour preoperatively in patients undergoing elective nephrectomy. Postoperatively, patients receive a patient controlled analgesia device for self delivering opioids. Morphine consumption in the first 48 hours is documented.

Hyperalgesia is measured by von-Frey-Filaments.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective nephrectomy

Exclusion Criteria:

* contraindication against pregabalin
* creatinine > 2.0 mg/dl
* GGT >165, AST >105, ALT >135
* peptic Ulcus
* haemorrhagic diathesis
* angina pectoris, myocardial infarction
* stroke
* bronchial asthma
* opioid abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Sandner-Kiesling, MD, Study Chair — Medical University of Graz; Helmar Bornemann-Cimenti, MD, DSc, Principal Investigator — Graz Medical University
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- See also: Medical University of Graz — http://www.medunigraz.at